CLINICAL TRIAL: NCT03714594
Title: A Randomized Study of the Effects of Dapagliflozin+Saxagliptin in Addition to Metformin Versus Single Addition Saxagliptin or Dapagliflozin on Glucose Metabolism in Patients With DM2 Poorly Controlled With Metformin
Brief Title: Effects of Dapagliflozin+Saxagliptin in Addition to Metformin v/s Saxagliptin or Dapagliflozin in Patients With DM2.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Prof. Stefano Del Prato, Clinical Resercher, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Saxa-Dapa 1
Record Dates: First submitted 2018-07-25; First posted 2018-10-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dapagliflozin 10mg (Active Comparator): Dapagliflozin inhibits SGLT2 promoting the excretion of glucose in the urine,and lowers the plasma glucose concentration. This class of drugs has been shown to effectively reduce the HbA1c at all stages of T2DM and can be used in combination of all other anti-diabetic agents including insulin.
  Interventions: Drug: Dapagliflozin 10mg
- Saxagliptin 5mg (Active Comparator): Saxagliptin is a DPP4 inhibitor.In patients with type 2 diabetes,administration of saxagliptin led to inhibition of DPP4 enzyme activity.After an oral glucose load,this DPP4 inhibition resulted in a increase in circulating levels of active incretin hormones include GLP-1 and GIP, decreased glucagon concentrations and increased glucose-dependent beta-cell responsiveness,which resulted in higher insulin and C-peptide concentrations.The rise in insulin from pancreatic beta-cells and the decrease in glucagon from pancreatic alpha-cells were associated with lower fasting glucose concentrations and reduced glucose excursion following an oral glucose load or a meal.Saxagliptin improves glycaemic control by reducing fasting and postprandial glucose concentrations in patients with type 2 diabetes.
  Interventions: Drug: Dapagliflozin 10mg; Drug: Saxagliptin 5mg
- Saxagliptin 5 mg + dapagliflozin 10 mg (Active Comparator): Please see Arm 1 and 2
  Interventions: Drug: Saxagliptin 5mg + Dapagliflozin 10 mg

INTERVENTIONS:
Drug: Dapagliflozin 10mg — Dapagliflozin inhibits subtype 2 of the sodium-glucose transport proteins (SGLT2) which are responsible for at least 90% of the glucose reabsorption in the kidney. Blocking this transporter mechanism causes blood glucose to be eliminated through the urine.[
  Other Names: forxiga
  Arms: Dapagliflozin 10mg; Saxagliptin 5mg
Drug: Saxagliptin 5mg — Inhibits DPP-4 and slows inactivation of incretin hormones, thereby increasing blood concentrations and reducing fasting and postprandial glucose concentrations in a glucose-dependent manner in patients with type 2 diabetes mellitus
  Other Names: Onglyza
  Arms: Saxagliptin 5mg
Drug: Saxagliptin 5mg + Dapagliflozin 10 mg — Please see Intervention 1 and 2
  Other Names: No other intervention name specified
  Arms: Saxagliptin 5 mg + dapagliflozin 10 mg

SUMMARY:
A phase IV, randomized, double-blind, single center pilot study in subjects with type 2 diabetes poorly controlled with metformin therapy will be randomized to receive, on top of metformin: saxagliptin (5 mg/day) and dapagliflozin (10 mg/day) (Group 1);saxagliptin (5 mg/day) and placebo (Group 2); dapagliflozin (10 mg/day) and placebo (Group 3) for 4 weeks.

DETAILED DESCRIPTION:
Dapagliflozin (Forxiga) currently is approved for the treatment of T2DM (6). Dapagliflozin inhibits SGLT2, promote the excretion of 80-90 grams of glucose per day in the urine, and lower the plasma glucose concentration. This class of drugs has been shown to effectively reduce the HbA1c at all stages of T2DM and can be used in combination of all other anti-diabetic agents including insulin.

Saxagliptin is a highly potent DPP4 inhibitor.In patients with type 2 diabetes, administration of saxagliptin led to inhibition of DPP4 enzyme activity for a 24-hour period.After an oral glucose load,this DPP4 inhibition resulted in a 2- to 3-fold increase in circulating levels of active incretin hormones, including glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), decreased glucagon concentrations and increased glucose-dependent beta-cell responsiveness, which resulted in higher insulin and C-peptide concentrations.The rise in insulin from pancreatic beta-cells and the decrease in glucagon from pancreatic alpha-cells were associated with lower fasting glucose concentrations and reduced glucose excursion following an oral glucose load or a meal.Saxagliptin improves glycaemic control by reducing fasting and postprandial glucose concentrations in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Age = 35-70 years
3. BMI ≤ 40 Kg/m 2 and stable weight (± 3 lbs) over the preceding three months
4. Type 2 diabetes (HbA1c > 7 % and < 10 %)
5. Metformin on stable dose (at least 1500 mg/day) for at least 12 weeks before screening and at study initiation.
6. Subjects who are women of childbearing potential must agree to utilize a highly effective contraceptive measure throughout the course of the study.. 7.7. Subjects are capable of giving informed consent

Exclusion Criteria:

1. Drugs known to affect glucose metabolism (other than metformin) for more than14 days during the 12 weeks before screening
2. Known Dapagliflozin and Saxagliptin Excipient Hypersensitivity
3. Type 1 Diabetes or History of Ketoacidosis
4. history of cancer of any type;
5. cerebrovascular or symptomatic peripheral vascular disease;
6. heart disease class III or IV NYHA;
7. Estimated glomerular filtration rate (eGFR) ≤60 mL/min/1.73m 2 or serum creatinine > 1.5mg/dL in men or >1.4mg/dL in women
8. Liver function enzymes higher more than two times the upper limit
9. Ongoing urinary tract infection
10. drug or alcohol abuse;
11. life expectancy <3 yrs
12. blood pressure >160/100 mmHg
13. Donation of blood to a blood bank, blood transfusion, or participation in a clinical study requiring withdrawal of > 400 mL of blood during the 8 weeks prior to the enrollment visit and at least 8 weeks thereafter
14. Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study (estrogen and/or progesterone treatment)
15. Women who are pregnant or breastfeeding
16. Patient with a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance which, in the opinion of the investigator or coordinator, might pose an unacceptable risk to the patient or interfere with trial procedures

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Glucose Metabolism | from first day
  To determine the effect of the combination of dapagliflozin (a SGLT2-inhibitor) and saxagliptin (a DPP-4 inhibitor) on pancreatic hormones secretion and endogenous glucose production in Type 2 diabetic subjects through comparison of the effects of co-administration of Saxagliptin and Dapagliflozin vs. Saxagliptin or Dapagliflozin alone.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Del prato, Principal Investigator — University of Pisa
Locations (1):
- Department of Endocrinology and Metabolism, University of Pisa, Pisa, Italy